CLINICAL TRIAL: NCT03334240
Title: A Phase 2, Randomized, Vehicle-controlled, Double-blind Study to Explore the Efficacy, Pharmacodynamics and Safety of Topical Ionic Contra-viral Therapy (ICVT) Comprised of Digoxin and Furosemide in HPV-induced Genital Lesions of Immunocompromised and Immunocompetent Patients
Brief Title: ICVT in HPV-induced Genital Lesions of Immunocompromised and Immunocompetent Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of effect in interim analysis
Sponsor: Maruho Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLS003-CO-PR-003
Record Dates: First submitted 2017-10-30; First posted 2017-11-07 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: HPV-Induced Genital Lesions
Keywords: HPV; Digoxin; Furosemide; Vulvar HSIL

STUDY DESIGN:
Intervention Model Description: A total of 48 subjects are planned to be enrolled within one of the following three groups: a.) Immunocompetent patients with anogenital warts, b.) Immunocompromised with anogenital warts and c.) Immunocompromised with vulvar HSIL [3:1, active/vehicle]. Eligible subjects may enroll in an (up to) 8-week open-label Part 2 of study
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- CLS003 (Experimental): Digoxin and Furosemide topical formulation
  Interventions: Drug: CLS003
- Vehicle (Placebo Comparator): Inactive vehicle
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: CLS003 — CLS003
  Arms: CLS003
Drug: Vehicle — Vehicle
  Arms: Vehicle

SUMMARY:
This study is intended to explore and evaluate the pharmacodynamics and clinical efficacy of the ionic contra-viral therapy CLS003 in immunocompromised and immunocompetent patients with benign and premalignant HPV-induced genital lesions

DETAILED DESCRIPTION:
This study is intended to explore clinical efficacy and safety/tolerability of ICVT as a potential treatment for benign and premalignant HPV-induced genital lesions in immunocompetent and immunosuppressed patients. This includes 3 different patient populations: i) immunocompetent patients with anogenital warts (AGWs), ii) immunocompromised patients with anogenital warts and iii) immunocompromised patients with vulvar high grade squamous intraepithelial neoplasia (HSIL), formerly referred to as usual type vulvar intraepithelial neoplasia (uVIN). Since digoxin / furosemide ICVT's mode of action is in part independent of the immune system and directly targeted to eradicate the causative HPV, we hypothesize this therapy to be of value in this specific group of individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years in general, stable good health (with the exception of the immunocompromised disorder) as per judgment of the investigator based upon the results of a medical history, physical examination, ECG, chemistry, hematology.
2. In case of immunocompromised patients including but not limited to; patients receiving immunosuppressive therapy for any reason, patients with auto-immune disease, HIV patients, transplantation patients
3. In case of genital warts patient group(s): have at least 3 genital warts (only applicable to Study Part 1)
4. In case of vulvar HSIL: at least one lesion that can be accurately measured in at least one dimension with longest diameter ≥ 20 mm OR in 2 perpendicular dimensions that when multiplied together give a surface area ≥ 120 mm² (only applicable to Study Part 1)
5. If female of childbearing potential, have a negative urine pregnancy test at Screening and Day 0, and is willing to use effective contraception during the study and 3 months afterwards (i.e. oral, implanted, injectable, IUD, diaphragm, condom, tubal ligation, abstinence, or are in a monogamous relationship with a partner who has had a vasectomy)
6. Able to participate and willing to give written informed consent and to comply with the study restrictions
7. Ability to communicate well with the investigator in the Dutch language
8. Willing to refrain from using other topical products in the treatment area, or prohibited medications for the duration of the study

Exclusion Criteria:

1. Significant, uncontrolled or unstable disease in any organ system as per judgment of the investigator (regardless of association with the immunosuppressing disorder/therapy), including but not limited to: psychiatric, neurologic, cardiovascular, pulmonary, gastrointestinal, hepatic, renal, endocrine, hematologic or respiratory disease
2. Have used or received any topical genital wart treatment, cryotherapy, electrocoagulation, surgery in the treatment area within 28 days prior to enrolment
3. Have used or received any topical vulvar HSIL treatment, laser therapy or surgery in the treatment area within 28 days prior to enrolment
4. Have any current relevant skin infections in the treatment area other than genital warts (inclusively, but not limited to atopic dermatitis, lichen sclerosis, lichen planus or psoriasis)
5. Have a known sensitivity to any of the investigational product ingredients, including digoxin and furosemide
6. Participation in an investigational drug or device study within 3 months prior to screening or more than 4 times in the past year
7. Loss or donation of blood over 500 mL within three months prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Lesion (vulvar HSIL or wart) size reduction | Day 0, 21, 42, 84, 126, (Part 1 of study), Day 0, 28, 56, 140 (Part 2 of study)
Change in patient-reported outcomes | Through study completion, up to 20 weeks
HPV viral load assessment | Day 0, 21, 42, 84, 126, (Part 1 of study), Day 0, 28, 56, 140 (Part 2 of study)
Change in the HPV viral load | Day 0, 21, 42, 84, 126, (Part 1 of study), Day 0, 28, 56, 140 (Part 2 of study)
Mean HPV viral load | Day 0, 21, 42, 84, 126, (Part 1 of study), Day 0, 28, 56, 140 (Part 2 of study)
Histology (regression of vulvar HSIL or AGWs to no dysplasia, HPV genotyping) | Day 0, 42, 126, (Part 1 of study), Day 56 (Part 2 of study)
Local immunity status | Day 0, 21, 42, 84, 126, (Part 1 of study), Day 0, 28, 56, 140 (Part 2 of study)
Percentage clearance of vulvar HSIL lesions | Day 0, 21, 42, 84, 126, (Part 1 of study), Day 0, 28, 56, 140 (Part 2 of study)
  For vulvar HSIL cohort
Proportion of patients with all vulvar HSIL lesions cleared | Day 0, 21, 42, 84, 126, (Part 1 of study), Day 0, 28, 56, 140 (Part 2 of study)
  For vulvar HSIL cohort
Histology (regression of vulvar HSIL to no dysplasia) | Day 0, 42, 126, (Part 1 of study), Day 56 (Part 2 of study)
  For vulvar HSIL cohort
Histological recurrence in the Part 1 follow-up period | Day 84, 126
  For vulvar HSIL cohort
Percentage clearance of genital warts | Day 0, 21, 42, 84, 126, (Part 1 of study), Day 0, 28, 56, 140 (Part 2 of study)
  For genital wart cohort
Proportion of patients with all genital warts cleared | Day 0, 21, 42, 84, 126, (Part 1 of study), Day 0, 28, 56, 140 (Part 2 of study)
  For genital wart cohort
Clinical recurrence in the Part 1 follow-up period | Day 84, 126
  For genital wart cohort

SECONDARY OUTCOMES:
Adverse event collection to assess safety/tolerability of CLS003 | Day 0, 21, 42, 84, 126, (Part 1 of study), Day 0, 28, 56, 140 (Part 2 of study), and as volunteered by patient

CONTACTS AND LOCATIONS:
Overall Officials: J. (Koos) Burggraaf, MD, PhD, Principal Investigator — Centre For Human Drug Research
Locations (1):
- LUMC/Centre For Human Drug Research, Leiden, Netherlands